CLINICAL TRIAL: NCT01058941
Title: Lipoic Acid and Omega-3 Fatty Acids in Alzheimer's Disease
Brief Title: Lipoic Acid and Omega-3 Fatty Acids for Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lynne Shinto, Lynne Shinto, ND, MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AG033613-01A1 (NIH)
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; fish oil; lipoic acid
MeSH Terms: conditions — Alzheimer Disease | interventions — Thioctic Acid; Fish Oils; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipoic acid and Omega-3 fatty acids (Experimental): Three 1-gram fish oil capsules per day (2 capsules in the morning and 1 capsule in the evening) plus two lipoic acid (LA) capsules per day in the morning. Total daily dose of study drug: 675 mg DHA, 975 mg EPA, 600 mg LA.
  Interventions: Drug: Lipoic acid and fish oil concentrate
- Placebo (Placebo Comparator): Three placebo oil capsules per day (2 capsules in the morning and 1 capsule in the evening) plus two placebo LA capsules per day in the morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lipoic acid and fish oil concentrate — Lipoic acid (600 milligrams per day) and fish oil concentrate (3 grams per day) for 18 months
  Other Names: alpha lipoic acid; thiotic acid; fish oil; omega-3 fatty acids
  Arms: Lipoic acid and Omega-3 fatty acids
Drug: Placebo — Placebo LA and placebo oil capsules for 18 months
  Other Names: Placebo for lipoic acid and fish oil concentrate
  Arms: Placebo

SUMMARY:
The purpose of this study was to see if taking lipoic acid plus omega-3 fatty acids (omega-3s) can slow the Alzheimer's disease (AD) process. To see if the treatment can slow the AD process, the investigators looked at changes in memory and changes in a person's daily activities over 18 months.

DETAILED DESCRIPTION:
Current pharmacological agents for AD have had no impact on disease prevalence and have had limited effects on improving the clinical course of AD. The exponential rise in the prevalence, incidence, and cost of care for AD make finding therapeutic agents that can either prevent AD or delay disease progression an urgent health care need. Since inflammation, lipid dysregulation, and insulin resistance have each been associated with AD pathology, the combination of lipoic acid plus fish oil has the potential to maximize therapeutic benefit by acting on all three mechanisms associated with disease pathology.

ELIGIBILITY:
Inclusion Criteria:

1. 55 years or older
2. Probable AD by National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association - NINCDS/ADRDA criteria
3. MMSE between 15-26
4. Caregiver/study partner that can accompany participant to all study visits
5. Stable use of cholinesterase inhibitors and memantine permitted - doses must be stable for 4 months prior to study enrollment
6. Stable doses of over-the-counter antioxidants (e.g. vitamin E, ginkgo biloba) are permitted - dose must be stable for 4 months prior to study enrollment
7. Stable dose of lipid lowering medication - dose must be stable for 4 months prior to study enrollment
8. Geriatric Depression Scale (GDS) - Score of < 5
9. General health status that will not interfere with the participant's ability to complete the study.
10. Screening laboratory values within normal limits or, if abnormal, deemed clinically insignificant by the investigator
11. Sufficient English language skills to complete all testing

Exclusion Criteria:

1. Non-AD dementia
2. Residence in nursing home facility at screening visit (residence in community assisted living and long-term care facilities in which the participant still performs majority of basic activities of daily living will not be an exclusion)
3. History of clinically significant stroke (stroke with neurologic deficits > 6 months after diagnosis)
4. Health conditions such as cancer diagnosed < 5 years prior to enrollment (prostate cancer gleason grade < 3 and non metastatic skin cancers are acceptable), liver disease, history of ventricular fibrillation or ventricular tachycardia, major psychiatric disorder, central nervous system diseases (e.g. brain tumor, seizure disorder)
5. Insulin dependent diabetes or uncontrolled diabetes (diabetes controlled on medications other than insulin are acceptable)
6. Hyperlipidemic (triglycerides >500 mg/dl, LDL > 160 mg/dl, total cholesterol >240 mg/dl). LDL levels between 160 mg/dl and 165 mg/dl will be reviewed by the PI and included if judged to be safe. Patients who have a history or hyperlipidemia, but are not taking lipid-lowering medications due to potential memory impairment side effects will be reviewed on a case-by-case basis by the PI and enrolled in the study if deemed safe by PI and the patient's primary care provider.
7. Fish intake of one 6 ounce serving > once a week less than 4 months prior to enrollment
8. Omega-3 fatty acid supplement intake (e.g. fish oil capsules, cod liver oil, or flaxseed oil) less than 4 months prior to enrollment
9. Lipoic Acid supplementation less than 1 month prior to enrollment
10. Taking systemic corticosteroids, neuroleptics, antiparkinsonian agents, and narcotic analgesics. Certain low dose antipsychotic use will be reviewed by the principle investigator on a case-by-case basis and may be allowed if determined that dose is not strong enough to affect performance on cognitive evaluations. Low dose sinemet and dopamine agonist taken once a day for restless leg syndrome is not an exclusion.
11. Contraindications to MRI (for subjects enrolled at Bend, Medford, and Klamath sites that decide not to undergo MRI, this will not be an exclusion).
12. Enrollment in another study

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Shinto, ND, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lipoic Acid and Omega-3 Fatty Acids: lipoic acid and fish oil concentrate
  lipoic acid and fish oil concentrate: lipic acid (600 milligrams per day) and fish oil concentrate (3 grams per day) for 18 months
- Placebo: placebo lipoic acid plus placebo oil
  lipoic acid and fish oil concentrate: lipic acid (600 milligrams per day) and fish oil concentrate (3 grams per day) for 18 months
Period: Overall Study
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
Started | 34 | 33
Completed | 25 | 22
Not Completed | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 29 | 29 | 58
Age, Continuous [Mean (Full Range); unit: years] | 73.3 [56 to 92] | 76.2 [52 to 89] | 74.7 [52 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 34 | 32 | 66
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 33 | 30 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Activities of Daily Living (ADL) at 18 Months
Description: The Alzheimer's Disease Cooperative Study Activities of Daily Living Scale (ADCS-ADL) is used to assess activities of daily living in people with AD using a structured interview to ask the AD participant's caregiver/study partner to assess functional ability over a wide range of performance measures. A higher ADL score indicates greater impairment in functional ability; scores range from 0 to 27.
Time Frame: Baseline and 18 months
Population: Twenty participants discontinued from the study prior to completing all study visits. One treatment participant did not complete the final ADL assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 24 | 22
units on a scale | -11.58 (12.68) | -13.45 (12.89)
Statistical Analysis 1: Comparison: Lipoic Acid and Omega-3 Fatty Acids vs Placebo; The target enrollment was 60 subjects, allowing for up to a 20% drop-out. It was calculated that with 48 subjects (24 per group) we would have 80% power to see differences in ADL scores over 18 months between the treatment and placebo groups with a significance level of 0.025 based on a simple Bonferroni adjustment, since we had two primary outcomes; Test type: Other; p = 0.82, Mixed Models Analysis — We used a significance level of p = 0.025 for our measure of ADL changes based on a simple Bonferroni adjustment since we have two primary outcomes; Adjusted for baseline outcome, time from baseline, age, education category, BMI, cholinesterase inhibitors, memantine, vitamin E, and Apo-E; Mean Difference (Net) = -0.42, 95% CI 2-sided [-3.97 to 3.13]

2. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog) at 18 Months
Description: The ADAS-cog assesses general cognitive function over multiple domains and evaluates memory, attention, reasoning, language, orientation, and praxis. A higher score indicates greater impairment on a range of scores from 0 to 70. A total score of 70 indicates maximum severity.
Time Frame: Baseline and 18 months
Population: Twenty participants discontinued from the study prior to completing all study visits. One placebo and one treatment participant did not complete the final ADAS-cog assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
Number analyzed (Participants) | 24 | 21
units on a scale | 6.61 (6.67) | 3.40 (4.50)
Statistical Analysis 1: Comparison: Lipoic Acid and Omega-3 Fatty Acids vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.001, Mixed Models Analysis — We used a significance level of p = 0.025 for our measure of ADAS-cog changes based on a simple Bonferroni adjustment since we have two primary outcomes; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -3.68, 95% CI 2-sided [-5.90 to -1.46]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored once a month as a part of the clinic visits and monthly by phone. Reported AEs include events that occurred on or after Day 0 and on or before month 18.
Arm/Group | Lipoic Acid and Omega-3 Fatty Acids | Placebo
All-Cause Mortality (participants affected / at risk) | 1/34 | 2/33
Serious Adverse Events (participants affected / at risk) | 10/34 | 7/33
Other Adverse Events (participants affected / at risk) | 29/34 | 27/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipoic Acid and Omega-3 Fatty Acids (N=34) | Placebo (N=33)
Drug-induced delirium (Psychiatric disorders) | 0 (0) | 1 (1) — Nyquil use
Dementia Alzheimer's Type (Nervous system disorders) | 2 (2) | 0 (0) — Rapid cognitive decline
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Fall down stairs
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subdural haematoma evacuation (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipoic Acid and Omega-3 Fatty Acids (N=34) | Placebo (N=33)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 7 (7)
Nausea (Gastrointestinal disorders) | 4 (6) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 7 (8)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (4)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (4)
Headache/Migraine (Nervous system disorders) | 5 (6) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Behavioral and psychiatric symptoms of dementia (Psychiatric disorders) | 4 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 4 (4) | 1 (1)
Allergic conditions (Immune system disorders) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 2 (3)
Sycope (Vascular disorders) | 2 (3) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No